CLINICAL TRIAL: NCT03815825
Title: A Phase 2, Randomized Placebo-Controlled, Double-Masked Study to Assess Safety and Efficacy of Multiple Doses of IONIS-FB-LRx, an Antisense Inhibitor of Complement Factor B, in Patients With Geographic Atrophy Secondary to Age-Related Macular Degeneration (AMD)
Brief Title: GOLDEN STUDY: A Study to Assess Safety and Efficacy of Multiple Doses of IONIS-FB-LRx in Participants With Geographic Atrophy Secondary to Age-Related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISIS 696844-CS5; 2020-005174-94 (EudraCT Number)
Record Dates: First submitted 2019-01-22; First posted 2019-01-24 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Macular Degeneration; Geographic Atrophy
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IONIS-FB-LRx (Experimental): Stage 1 participants will receive IONIS-FB-LRx randomized to 1 of 3 dose levels, administered subcutaneously every 4 weeks, completing the treatment period at Week 45. Stage 2 will expand 2 of the dosing cohorts in a new randomized group of participants based on the Stage 1 interim analysis. Participants will be randomized to 1 of 2 of the expanded cohorts, administered subcutaneously every 4 weeks, completing the treatment period at Week 45.
  Interventions: Drug: IONIS-FB-LRx
- Placebo (Experimental): Stage 1 participants will receive a placebo matching solution, administered subcutaneously every 4 weeks, completing the treatment period at Week 45. Stage 2 participants will receive a placebo matching solution, administered subcutaneously every 4 weeks, completing the treatment period at Week 45.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IONIS-FB-LRx — IONIS-FB-LRx at multiple ascending doses, administered subcutaneously every 4 weeks
  Other Names: ISIS 696844
  Arms: IONIS-FB-LRx
Drug: Placebo — Placebo matching solution, administered subcutaneously every 4 weeks
  Arms: Placebo

SUMMARY:
Evaluate the effect of IONIS-FB-LRx on the rate of change of the area of geographic atrophy (GA) secondary to age-related macular degeneration (AMD) measured by fundus autofluorescence (FAF).

DETAILED DESCRIPTION:
The study will assess the rate of change of the area of GA secondary to AMD by measuring FAF in up to 330 participants with GA due to AMD being treated with IONIS-FB-LRx. The study is a Phase 2, double-masked, randomized, stratified, placebo-controlled study conducted at multiple centers. It is an adaptive design in which three dose levels will be evaluated in a subset of participants (Stage 1) and, following an interim analysis, the number of participants in two of the dose cohorts will be expanded (Stage 2).

ELIGIBILITY:
Inclusion Criteria:

* Females must be non-pregnant and non-lactating, and either surgically sterile or post-menopausal.
* Vaccination against Neisseria meningitidis and Streptococcus pneumoniae received at least 2 weeks prior to first dose of investigational product
* Well-demarcated geographic atrophy (GA) due to AMD
* Best-corrected visual acuity (BCVA) letter score of 35 letters (approx. 20/200 Snellen equivalent) or better on the ETDRS chart
* Must have clear ocular media and adequate pupillary dilation in the study eye to permit high-quality fundus imaging

Exclusion Criteria:

* Clinically-significant abnormalities in medical history
* A lack of full recovery from any infection for at least 14 days prior to the Study Drug administration
* Chronic treatment with steroids, including topically or intravitreally administered
* History or presence of diabetic retinopathy or diabetic macular edema (DME)
* History or presence of a disease other than AMD that could affect vision or safety assessments
* Prior treatment with another investigational drug, biological agent, or device
* Other protocol-specified inclusion/exclusion criteria may apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Rate of Change from Baseline in the Geographic Atrophy (GA) Area at Week 49, as Assessed by Retinal Imaging | Week 49

SECONDARY OUTCOMES:
Absolute change in the GA area from Baseline as measured by Fundus Autofluorescence (FAF) | Baseline and up to Week 57
Percentage Change from Baseline in Levels of Factor B (FB) in Plasma | Baseline and up to Week 49
Percentage Change from Baseline in Levels of Serum AH50 Activity | Baseline and up to Week 49
Absolute Change from Baseline in Low Luminance Visual Acuity (LLVA) | Baseline and up to Week 49

CONTACTS AND LOCATIONS:
Locations (80):
- United States (50):
  - IONIS Investigative Site, Phoenix, Arizona
  - IONIS Investigative Site, Sun City, Arizona
  - IONIS Investigative Site, Beverly Hills, California
  - IONIS Investigative Site, Huntington Beach, California
  - IONIS Investigative Site, La Jolla, California
  - IONIS Investigative Site, Long Beach, California
  - IONIS Investigative Site, Poway, California
  - IONIS Investigative Site, San Francisco, California
  - IONIS Investigative Site, Colorado Springs, Colorado
  - IONIS Investigative Site, Clearwater, Florida
  - IONIS Investigative Site, Fort Myers, Florida
  - IONIS Investigative Site, Lake Worth, Florida
  - IONIS Investigative Site, Lakeland, Florida
  - IONIS Investigative Site, Melbourne, Florida
  - IONIS Investigative Site, Stuart, Florida
  - IONIS Investigative Site, Tampa, Florida
  - IONIS Investigative Site, Winter Haven, Florida
  - IONIS Investigative Site, Augusta, Georgia
  - IONIS Investigative Site, Lemont, Illinois
  - IONIS Investigative Site, Springfield, Illinois
  - IONIS Investigative Site, Leawood, Kansas
  - IONIS Investigative Site, Baltimore, Maryland
  - IONIS Investigative Site, Hagerstown, Maryland
  - IONIS Investigative Site, Southaven, Mississippi
  - IONIS Investigative Site, Albuquerque, New Mexico
  - IONIS Investigative Site, Asheville, North Carolina
  - IONIS Investigative Site, Hickory, North Carolina
  - IONIS Investigative Site, Winston-Salem, North Carolina
  - IONIS Investigative Site, Cleveland, Ohio
  - IONIS Investigative Site, Tulsa, Oklahoma
  - IONIS Investigative Site, Philadelphia, Pennsylvania
  - IONIS Investigative Site, Pittsburgh, Pennsylvania
  - IONIS Investigative Site, West Mifflin, Pennsylvania
  - IONIS Investigative Site, Greenville, South Carolina
  - IONIS Investigative Site, Ladson, South Carolina
  - IONIS Investigative Site, Nashville, Tennessee
  - IONIS Investigative Site, Abilene, Texas
  - IONIS Investigative Site, Arlington, Texas
  - IONIS Investigative Site, Austin, Texas
  - IONIS Investigative Site, Bellaire, Texas
  - IONIS Investigative Site, Dallas, Texas
  - IONIS Investigative Site, McAllen, Texas
  - IONIS Investigative Site, San Antonio, Texas
  - IONIS Investigative Site, Southlake, Texas
  - IONIS Investigative Site, The Woodlands, Texas
  - IONIS Investigative Site, Willow Park, Texas
  - IONIS Investigative Site, Salt Lake City, Utah
  - IONIS Investigative Site, Lynchburg, Virginia
  - IONIS Investigative Site, Richmond, Virginia
  - IONIS Investigative Site, Silverdale, Washington
- Australia (11):
  - IONIS Investigative Site, Albury, New South Wales
  - IONIS Investigative Site, Hurstville, New South Wales
  - IONIS Investigative Site, Parramatta, New South Wales
  - IONIS Investigative Site, Sydney, New South Wales
  - IONIS Investigative Site, Adelaide, South Australia
  - IONIS Investigative Site, East Melbourne, Victoria
  - IONIS Investigative Site, Essendon, Victoria
  - IONIS Investigative Site, Glen Iris, Victoria
  - IONIS Investigative Site, Malvern, Victoria
  - IONIS Investigative Site, Parkville, Victoria
  - IONIS Investigative Site, Perth, Western Australia
- Austria (3):
  - IONIS Investigative Site, Linz, Upper Austria
  - IONIS Investigative Site, Klagenfurt
  - IONIS Investigative Site, Vienna
- Canada (3):
  - IONIS Investigative Site, London, Ontario
  - IONIS Investigative Site, Ottawa, Ontario
  - IONIS Investigative Site, Québec, Quebec
- IONIS Investigative Site, Prague, Czechia
- Netherlands (2):
  - IONIS Investigative Site, Nijmegen, Gelderland
  - IONIS Investigative Site, Rotterdam
- IONIS Investigative Site, Christchurch, New Zealand
- Poland (2):
  - IONIS Investigative Site, Katowice, Silesian
  - IONIS Investigative Site, Bydgoszcz
- Spain (7):
  - IONIS Investigative Site, Terrassa, Barcelona
  - IONIS Investigative Site, Majadahonda, Madrid
  - IONIS Investigative Site, Pamplona, Navarre
  - IONIS Investigative Site, Burjassot, Valencia
  - IONIS Investigative Site, Barcelona
  - IONIS Investigative Site, Valladolid
  - IONIS Investigative Site, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tzoumas N, Riding G, Williams MA, Steel DH. Complement inhibitors for age-related macular degeneration. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD009300. doi: 10.1002/14651858.CD009300.pub3. PMID 37314061